CLINICAL TRIAL: NCT02790853
Title: Multimodal Imaging for Surveillance of Patients With Oral Potentially Malignant Disorders
Brief Title: Multimodal Imaging for Surveillance in Patients With Oral Potentially Malignant Disorders
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-0831; NCI-2018-02554 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0831 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2016-05-26; First posted 2016-06-06 (Estimated); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Dysplasia; Lip and Oral Cavity Carcinoma; Oral Disorder; Premalignant Lesion
MeSH Terms: conditions — Mouth Neoplasms; Mouth Diseases | interventions — Biopsy; Optical Imaging; Proflavine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Diagnostic (multimodal imaging, biopsy) (Experimental): Participants undergo PS2.1/PS3 imaging and high-resolution microendoscope imaging with proflavine hemisulfate applied to the mucosa. Patients also undergo brush biopsy and incisional biopsy. Procedures are repeated every 3-4 months for 2 years.
  Interventions: Procedure: Biopsy; Procedure: Fluorescence Imaging; Procedure: High-Resolution Microendoscopy; Drug: Proflavine Hemisulfate

INTERVENTIONS:
Procedure: Biopsy — Undergo brush biopsy and incisional biopsy
  Other Names: Bx
Procedure: Fluorescence Imaging — Undergo PS2.1/PS3 imaging
Procedure: High-Resolution Microendoscopy — Undergo HRME imaging
  Other Names: HRME
Drug: Proflavine Hemisulfate — Applied on mucosa

SUMMARY:
This early phase I trial studies how well multimodal imaging works for surveillance in patients with oral potentially malignant disorders. New types of imaging devices may help doctors decide if a lesion in the mouth is pre-cancerous or cancerous.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare standard white light examination to multimodal imaging for detection of high grade dysplasia and carcinoma during follow-up examinations of patients with oral potentially malignant disorders (OPMD).

SECONDARY OBJECTIVES:

I. To determine qualitative and quantitative diagnostic assessment of patients who agree to undergo imaging and have images of sufficient quality.

II. To compare expression of molecular biomarkers to results from white light examination, multimodal imaging and pathologic assessment in a subset of patients who have invasive biopsies or resection.

III. To compare cytologic results from brush biopsy specimens to white light examination and multimodal imaging results.

OUTLINE:

Participants undergo PS2.1/PS3 imaging and high-resolution microendoscope imaging with proflavine hemisulfate applied to the mucosa. Patients also undergo brush biopsy and incisional biopsy. Procedures are repeated every 3-4 months for 2 years.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are willing to participate.
* Adult subjects with: a. clinically evident oral premalignant lesion (OPL) or suspicious oral mucosal lesion. or b. pathologic diagnosis of dysplasia or c. history of resected oral cancer or d. oral potentially malignant disorder (OPMD) or e. history of tobacco and/or alcohol exposure.
* Ability to understand and willingness to sign a written informed consent document (ICD).

Exclusion Criteria:

* Known allergy to proflavine or acriflavine.
* Pregnant females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-05-25 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Detection of high grade dysplasia and carcinoma | Up to 2 years
  Will compare standard white light examination to multimodal imaging for detection of high grade dysplasia and carcinoma during follow-up examinations of patients with oral potentially malignant disorders (OPMD).

SECONDARY OUTCOMES:
Diagnostic assessment | Up to 2 years
  Will determine qualitative and quantitative diagnostic assessment of patients who agree to undergo imaging and have images of sufficient quality.
Biomarker analysis | Up to 2 years
  Will compare expression of molecular biomarkers to results from white light examination, multimodal imaging and pathologic assessment in a subset of patients who have invasive biopsies or resection.
Cytologic results | Up to 2 years
  Will compare cytologic results from brush biopsy specimens to white light examination and multimodal imaging results.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Gillenwater, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org